CLINICAL TRIAL: NCT06664476
Title: The Effect of Educational Program on Nurses' Knowledge and Practice Regarding Implanted Port-A-Catheter Care for Patients Undergoing Chemotherapy
Brief Title: Educational Program's Impact on Nurses' Skills in Port-A-Catheter Care for Chemotherapy Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohammed Elsayed Zaky, Principal Investigator, Cairo University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Nurses' Knowledge and Practice
Record Dates: First submitted 2024-10-25; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Chemotherapy
Keywords: Implanted Port-A-Catheter; Oncology Nursing; Chemotherapeutic Management; Nurses' Knowledge

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): The study group for this research consists of 45 oncology nurses who are actively involved in the care and management of patients with implanted Port-A-Catheters for chemotherapy. These nurses are recruited from the Oncology and Nuclear Medicine Center at Kasr Elini hospital, which includes outpatient clinics. The nurses in this study play a critical role in handling long-term venous access devices, particularly Port-A-Catheters, which are essential for the administration of chemotherapy and other related treatments.
  Interventions: Behavioral: PortCare Professional Training Program

INTERVENTIONS:
Behavioral: PortCare Professional Training Program — The intervention is a targeted educational program to enhance oncology nurses' skills in managing Port-A-Catheters for chemotherapy patients. It includes a preparatory phase to assess baseline knowledge and practices, followed by an implementation phase with theoretical and practical training. Theoretical sessions cover device basics and care guidelines, while practical sessions provide hands-on training on procedures like catheter insertion, flushing, and removal. This program aims to improve patient safety, reduce complications, and boost nurses' confidence in Port-A-Catheter care.

SUMMARY:
The goal of this experimental study is to evaluate if an educational intervention can improve nurses' knowledge and practice in caring for patients with implanted Port-A-Catheters among oncology nurses directly involved in chemotherapy care. The main questions it aims to answer are:

Will the educational program improve nurses' knowledge regarding Port-A-Catheter care? Will the educational program positively impact nurses' practical skills and reduce complications related to Port-A-Catheter management? Researchers will compare pre-intervention and post-intervention performance to see if the educational program leads to better knowledge and practice outcomes.

Participants will:

Attend a theoretical training session on Port-A-Catheter fundamentals, including its use, benefits, and common complications.

Engage in a practical session, involving demonstrations and supervised practice of Port-A-Catheter care, such as insertion, flushing, and removal.

Be evaluated before the intervention, immediately after, and at 2 weeks post-intervention to assess improvements and retention of knowledge and skills.

DETAILED DESCRIPTION:
Cancer is a rapidly growing, invasive, and metastatic disease caused by an accumulation of genetic mutations that lead to the formation of malignant cells. These genetic changes can result from exposure to chemical carcinogens, chronic inflammation, radiation, or a genetic predisposition. Globally, cancer is a significant public health challenge and ranks as the second leading cause of death in the United States. In recent years, the global burden of cancer has surged, with millions of new cases and fatalities each year. In Egypt, the numbers reflect a similar pattern, highlighting the widespread impact of this disease.

Chemotherapy remains the most commonly used treatment for cancer, utilizing chemical agents that target and destroy cancer cells, preventing their growth and spread. Often, chemotherapy is combined with other treatment modalities like surgery or radiation. While chemotherapy can be delivered through various routes, intravenous (IV) administration is the most common. Modern chemotherapy management requires consistent and safe access to the venous system for the delivery of drugs, fluids, and blood products. Due to the damaging effects of repeated venipuncture and long-term chemotherapy on peripheral veins, long-term venous access devices (VADs) have become essential. One of the most frequently used VADs is the Port-A-Catheter system.

A Port-A-Catheter is a medical device that provides direct access to large blood vessels. It consists of a reservoir (or portal) and a catheter, implanted in a surgically created pocket on the chest wall or upper arm. The portal is placed subcutaneously and connects to the catheter with a specialized lock. It can be used for chemotherapy 12 to 24 hours after insertion and typically remains in place for two to six years.

This device significantly reduces the pain and anxiety associated with repeated needle sticks or venous procedures, allowing patients greater freedom and safety in their daily activities. The Port-A-Catheter enables the delivery of chemotherapy agents, blood products, parenteral nutrition, and the collection of blood samples for testing, all contributing to an improved quality of life.

The primary benefits of ports include easier venous access, especially for patients with small or compromised veins, a lower risk of chemotherapy extravasation, and the ability to administer irritating substances. However, Port-A-Catheters are not without risks, which are categorized as early or delayed complications. Early complications may involve incorrect catheter positioning, pneumothorax, hemothorax, thoracic duct injury, or cardiac tamponade. Delayed complications include infections, thrombosis, stenosis, catheter fractures, and migration.

Proper nursing care and maintenance of implanted ports are crucial to keeping them functional and preventing complications. This care includes regular flushing, heparin locking, dressing changes, needle replacements, and scrubbing the access port with antiseptic solutions to minimize contamination risks. Nurses play a pivotal role in maintaining the integrity of the port, preventing failure, and reducing complications related to its use. Effective nursing care requires sharp assessment skills and sound clinical judgment to identify and manage central venous access device (CVAD) complications effectively.

ELIGIBILITY:
Inclusion Criteria:

* Nurses with at least one year of experience in oncology or chemotherapy units.
* Nurses currently working in the Oncology Care Center or related units that handle Port-A-Catheters.

Exclusion Criteria:

* Staff nurses working with experience less than least 6 months.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-10-29 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Nurses' knowledge regarding implanted port-A-Catheter care for patients undergoing Chemotherapy "Structured Interview Questionnaire | 2 weeks
  This part will be concerning with assessing nurses' knowledge about implanted port -A Catheter care for patients undergoing chemotherapy. It will include "thirty-eight" multiple choice questions; which will cover the following: "ten" questions are in relation to "General Nurses' knowledge about implanted port -A-Catheter", fourteen questions are about "Catheter connection and disconnection nursing care", "three" questions concerning "Catheter exit site care", "two" questions regarding "Port-A Catheter removal, "one" question about "patient documentation" and "eight" questions related to "Port-A-Catheter infection and complications".

SECONDARY OUTCOMES:
Oncology Nurses' Practices regarding Implanted Port-A-Catheter Care for Patients undergoing Chemotherapy Observational Checklist | 2 week
  Used to assess nurse's practice for port catheter (Accessing/ De-accessing, flushing, and removal of the noncoring safety needle of implanted port catheter).
  Each item will be checked as: "Done correctly" took "One" score and "Not done" or "Incorrectly done" had "Zero", with a total score of "117" grades. The total nurses' practices score will be calculated and transferred to percentage reflecting the levels of practices as follows: "Less than 60%" are considered "Poor practice level" "From 60% -75 %" reflects "Fair practice level" "More than 75%" denotes "Good practice level"

CONTACTS AND LOCATIONS:
Locations (1):
- Faculy of Nursing Kafr El sheikh University, Cairo, Egypt

REFERENCES:
- [Result] Mohamed, S., Talaat, E., & Falts, S. (2019). Assess nurses' performance regarding care of patient with implanted port undergoing chemotherapy. Egyptian Journal of Health C Alzuhairy, B. I. J., Al Zobair, A. A., & Al-Faqe, F. M. M. (2021). Complications of Port-A-Cath use for chemotherapy, drugs, and fluid administration in Mosul city. Archivos Venezolanos de Farmacología y Terapéutica, 40(4), 377-383
- [Result] Rossi F, Noren H, Jove R, Beljanski V, Grinnemo KH. Differences and similarities between cancer and somatic stem cells: therapeutic implications. Stem Cell Res Ther. 2020 Nov 18;11(1):489. doi: 10.1186/s13287-020-02018-6. PMID 33208173